CLINICAL TRIAL: NCT05061693
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study of the Efficacy and Safety of INCB054707 in Participants With Prurigo Nodularis
Brief Title: A Study to Evaluate the Efficacy and Safety of INCB054707 in Participants With Prurigo Nodularis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 54707-206; 2021-006329-23 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo nodularis; PN; INCB054707; chronic pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INCB054707 Dose A (Experimental): Participants will receive INCB054707 Dose A for 16 weeks (Period 1), followed by INCB054707 Dose B (responders) or by INCB054707 Dose C (partial or nonresponders) for 24 weeks (Period 2).
  Interventions: Drug: INCB054707
- INCB054707 Dose B (Experimental): Participants will receive INCB054707 Dose B for 16 weeks (Period 1), followed by INCB054707 Dose B (responders) or by INCB054707 Dose C (partial or nonresponders) for 24 weeks (Period 2).
  Interventions: Drug: INCB054707
- INCB054707 Dose C (Experimental): Participants will receive INCB054707 Dose C for 16 weeks (Period 1), followed by INCB054707 Dose B (responders) or by INCB054707 Dose C (partial or nonresponders) for 24 weeks (Period 2).
  Interventions: Drug: INCB054707
- Placebo followed by INCB054707 Dose B or C (Placebo Comparator): Participants will receive placebo for 16 weeks (Period 1), followed by INCB054707 Dose B (responders) or by INCB054707 Dose C (partial or nonresponders) for 24 weeks (Period 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB054707 — Oral; Tablet
  Other Names: Povorcitinib
  Arms: INCB054707 Dose A; INCB054707 Dose B; INCB054707 Dose C
Drug: Placebo — Oral; Tablet
  Arms: Placebo followed by INCB054707 Dose B or C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of INCB054707 in participants with prurigo nodularis over a 16-week double-blind placebo-controlled treatment period, followed by a 24 -week single blind extension period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PN for at least 3 months before screening.
* Inadequate response or intolerant to ongoing or prior PN therapy.
* ≥ 20 pruriginous lesions on ≥ 2 different body regions at screening and Day 1.
* Willingness to avoid pregnancy or fathering children
* Further inclusion criteria apply.

Exclusion Criteria:

* Have chronic pruritus due to a condition other than PN; have neuropathic and psychogenic pruritus such as but not limited to notalgia paresthetica, brachioradial pruritus, small fiber neuropathy, skin picking syndrome, or delusional parasitosis.
* Current use of a medication known to cause pruritus.
* Women who are pregnant (or who are considering pregnancy) or lactating.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q-wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis.
* Participants known to be infected with HIV, Hepatitis B, or Hepatitis C.
* Laboratory values outside of the protocol-defined ranges.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (49):
- United States (23):
  - Investigative Site US010, Phoenix, Arizona
  - Investigative Site US024, Phoenix, Arizona
  - Investigative Site US001, Fountain Valley, California
  - Investigative Site US014, Sacramento, California
  - Investigative Site US019, Fort Lauderdale, Florida
  - Investigative Site US016, Miami, Florida
  - Investigative Site US013, Miramar, Florida
  - Investigative Site US009, Tampa, Florida
  - Investigative Site 1071320, Newnan, Georgia
  - Investigative Site US008, Plainfield, Indiana
  - Investigative Site US011, South Bend, Indiana
  - Investigative Site US003, Baltimore, Maryland
  - Investigative Site US017, Troy, Michigan
  - Investigative Site US006, Saint Joseph, Missouri
  - Investigative Site US004, Portsmouth, New Hampshire
  - Investigative Site US023, Athens, Ohio
  - Investigative Site US002, Dublin, Ohio
  - Investigative Site US012, Gahanna, Ohio
  - Investigative Site US022, Murfreesboro, Tennessee
  - Investigative Site US021, Arlington, Texas
  - Investigative Site US005, Austin, Texas
  - Investigative Site US018, Dallas, Texas
  - Investigative Site US007, Houston, Texas
- Canada (4):
  - Investigative Site CA002, Edmonton, Alberta
  - Investigative Site CA001, Surrey, British Columbia
  - Investigative Site CA004, London, Ontario
  - Investigative Site CA003, Québec, Quebec
- Germany (7):
  - Investigative Site DE007, Bad Bentheim
  - Investigative Site DE005, Berlin
  - Investigative Site DE004, Bonn
  - Investigative Site DE003, Frankfurt am Main
  - Investigative Site DE001, Hamburg
  - Investigative Site DE002, Münster
  - Investigative Site DE008, Tübingen
- Poland (5):
  - Investigative Site PL005, Kielce
  - Investigative Site PL003, Osielsko
  - Investigative Site PL001, Rzeszów
  - Investigative Site PL004, Torun
  - Investigative Site PL002, Wroclaw
- Puerto Rico (2):
  - Investigative Site PR002, Caguas
  - Investigative Site PR001, San Juan
- Spain (8):
  - Investigative Site ES004, Alicante
  - Investigative Site ES007, Badalona
  - Investigative Site ES001, Barcelona
  - Investigative Site ES002, Córdoba
  - Investigative Site ES006, Granada
  - Investigative Site ES008, Madrid
  - Investigative Site ES003, Madrid
  - Investigative Site ES005, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted across 40 sites in Canada, Germany, Spain, Poland, Puerto Rico, and the United States.
Groups:
- PC Period: Placebo: On Day 1, participants were randomized to receive matching placebo once daily (QD) and stratified by Investigator's Global Assessment (IGA) score (3 versus 4). Participants received blinded study drug through Week 16.
- PC Period: Povorcitinib 15 mg: On Day 1, participants were randomized to receive povorcitinib 15 milligrams (mg) QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- PC Period: Povorcitinib 45 mg: On Day 1, participants were randomized to receive povorcitinib 45 mg QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- PC Period: Povorcitinib 75 mg: On Day 1, participants were randomized to receive povorcitinib 75 mg QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- Extension Period: Placebo to Povorcitinib 45 mg: Participants who received placebo during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch Numerical Rating Scale (NRS) score and Investigator's Global Assessment-Treatment Success (IGA-TS) who did not receive rescue therapy during the placebo-controlled period.
- Extension Period: Povorcitinib 15 mg to 45 mg: Participants who received povorcitinib 15 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Extension Period: Povorcitinib 45 mg to 45 mg: Participants who received povorcitinib 45 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for an additional 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Extension Period: Povorcitinib 75 mg to 45 mg: Participants who received povorcitinib 75 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Extension Period: Placebo to Povorcitinib 75 mg: Participants who received placebo during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Extension Period: Povorcitinib 15 mg to 75 mg: Participants who received povorcitinib 15 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Extension Period: Povorcitinib 45 mg to 75 mg: Participants who received povorcitinib 45 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Extension Period: Povorcitinib 75 mg to 75 mg: Participants who received povorcitinib 75 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for an additional 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
Period: 16-week Placebo-controlled (PC) Period
Arm/Group | PC Period: Placebo | PC Period: Povorcitinib 15 mg | PC Period: Povorcitinib 45 mg | PC Period: Povorcitinib 75 mg | Extension Period: Placebo to Povorcitinib 45 mg | Extension Period: Povorcitinib 15 mg to 45 mg | Extension Period: Povorcitinib 45 mg to 45 mg | Extension Period: Povorcitinib 75 mg to 45 mg | Extension Period: Placebo to Povorcitinib 75 mg | Extension Period: Povorcitinib 15 mg to 75 mg | Extension Period: Povorcitinib 45 mg to 75 mg | Extension Period: Povorcitinib 75 mg to 75 mg
Started | 37 | 36 | 36 | 37 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 32 | 29 | 31 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 7 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 24-week Extension Period
Arm/Group | PC Period: Placebo | PC Period: Povorcitinib 15 mg | PC Period: Povorcitinib 45 mg | PC Period: Povorcitinib 75 mg | Extension Period: Placebo to Povorcitinib 45 mg | Extension Period: Povorcitinib 15 mg to 45 mg | Extension Period: Povorcitinib 45 mg to 45 mg | Extension Period: Povorcitinib 75 mg to 45 mg | Extension Period: Placebo to Povorcitinib 75 mg | Extension Period: Povorcitinib 15 mg to 75 mg | Extension Period: Povorcitinib 45 mg to 75 mg | Extension Period: Povorcitinib 75 mg to 75 mg
Started | 0 | 0 | 0 | 0 | 1 | 4 | 8 | 15 | 30 | 25 | 23 | 18
Completed | 0 | 0 | 0 | 0 | 1 | 4 | 7 | 12 | 25 | 22 | 18 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 3 | 5 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Site Closure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: On Day 1, participants were randomized to receive matching placebo once daily (QD) and stratified by Investigator's Global Assessment (IGA) score (3 versus 4). Participants received blinded study drug through Week 16.
- Povorcitinib 15 mg: On Day 1, participants were randomized to receive povorcitinib 15 milligrams (mg) QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- Povorcitinib 45 mg: On Day 1, participants were randomized to receive povorcitinib 45 mg QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- Povorcitinib 75 mg: On Day 1, participants were randomized to receive povorcitinib 75 mg QD and stratified by IGA score (3 versus 4). Participants received blinded study drug through Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg | Total
Number analyzed (Participants) | 37 | 36 | 36 | 37 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (12.32) | 56.0 (12.92) | 55.6 (15.25) | 55.9 (10.18) | 55.1 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 27 | 23 | 96
  Male | 15 | 12 | 9 | 14 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 3 | 3 | 16
  Not Hispanic or Latino | 30 | 32 | 33 | 33 | 128
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 33 | 31 | 27 | 30 | 121
  Black/African-American | 3 | 3 | 5 | 5 | 16
  Asian | 0 | 2 | 4 | 1 | 7
  American-Indian/Alaska Native | 0 | 0 | 0 | 1 | 1
  Unknown | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥4-point Improvement in Itch Numerical Rating Scale (NRS) Score at Week 16
Description: Each evening, the participants assessed their worst level of itch during the past 24 hours on a scale of 0 (no itch) to 10 (worst itch imaginable). The Baseline Itch NRS score was determined by averaging the 7 daily Itch NRS scores before Day 1 (i.e., Day -7 to Day -1). If ≥4 of the 7 days of the daily Itch NRS scores were missing prior to Day 1, then the Baseline Itch NRS score was set to "missing." The by-visit Itch NRS score for postbaseline visits was determined by averaging the 7 daily Itch NRS scores before the visit day. If 4 or more daily Itch NRS scores out of the 7 days before the visit day were missing, the Itch NRS score at the visit was set to missing.
Time Frame: Baseline; Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups for this population were defined according to the treatment assignment at randomization. Missing post-Baseline values and rescue therapy recipients for all subsequent visits after the initiation date of rescue therapy were imputed as nonresponders. The 95% confidence interval was based on the Clopper-Pearson exact method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 37 | 36 | 36 | 37
percentage of participants | 8.1 [1.7 to 21.9] | 36.1 [20.8 to 53.8] | 44.4 [27.9 to 61.9] | 56.8 [39.5 to 72.9]
Statistical Analysis 1: Comparison: Placebo vs Povorcitinib 15 mg; Test type: Superiority; p = 0.0061, Regression, Logistic; Exact Logistic regression: (response at Week 16 = treatment + stratification factor [Day 1 Investigator's Global Assessment score (3 or 4)]); Odds Ratio (OR) = 7.1, 95% CI 2-sided [1.6 to 45.4]
Statistical Analysis 2: Comparison: Placebo vs Povorcitinib 15 mg; Test type: Superiority; difference in response rate = 28.0, Standard Error of Mean 9.18 — The standard error of the difference between response rates was from normal approximation
Statistical Analysis 3: Comparison: Placebo vs Povorcitinib 45 mg; Test type: Superiority; p = 0.0005, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 10.2, 95% CI 2-sided [2.3 to 65.6]
Statistical Analysis 4: Comparison: Placebo vs Povorcitinib 45 mg; Test type: Superiority; difference in response rate = 36.3, Standard Error of Mean 9.42 — The standard error of the difference between response rates was from normal approximation
Statistical Analysis 5: Comparison: Placebo vs Povorcitinib 75 mg; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 16.8, 95% CI 2-sided [3.9 to 107.5]
Statistical Analysis 6: Comparison: Placebo vs Povorcitinib 75 mg; Test type: Superiority; difference in response rate = 48.6, Standard Error of Mean 9.30 — The standard error of the difference between response rates was from normal approximation

2. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment-Treatment Success (IGA-TS) (IGA Score of 0 or 1 With a ≥2-grade Improvement From Baseline) at Week 16
Description: The IGA for chronic prurigo considers the number of pruriginous lesions, which includes papules, nodules, plaques, umbilicated ulcers, and ulcers, and uses them as an overall severity rating on a scale of 0 to 4. 0: clear; no pruriginous lesions (0 lesions). 1: almost clear; rare palpable pruriginous lesions (approximately 1-5 lesions). 2: mild; few palpable pruriginous lesions (approximately 6-19 lesions). 3: moderate: many palpable pruriginous lesions (approximately 20-100 lesions). 4: severe; abundant palpable pruriginous lesions (over 100 lesions). The IGA-TS is defined as an IGA score of 0 or 1 with a ≥2-grade improvement from Baseline.
Time Frame: Baseline; Week 16
Population: ITT Population. Missing post-Baseline values were imputed as non-responders. The 95% confidence interval was based on the Clopper-Pearson exact method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 37 | 36 | 36 | 37
percentage of participants | 5.4 [0.7 to 18.2] | 13.9 [4.7 to 29.5] | 30.6 [16.3 to 48.1] | 48.6 [31.9 to 65.6]

3. Secondary Outcome: Time to ≥4-point Improvement From Baseline in Itch NRS Score
Description: as for outcome 1
Time Frame: up to 122 days
Population: ITT Population. The time to a ≥4-point improvement from Baseline in itch NRS score was estimated using the Kaplan-Meier method. The confidence interval for the median time to a ≥4-point improvement from Baseline was calculated using the method of Brookmeyer and Crowley. Only participants with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 36 | 35 | 34 | 36
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a ≥4-point improvement from Baseline in itch NRS score. | 58.0 [16.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a ≥4-point improvement from Baseline in itch NRS score. | 35.0 [21.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a ≥4-point improvement from Baseline in itch NRS score. | 19.0 [13.0 to 47.0]

4. Secondary Outcome: PC Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE is any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug up to 30 days after the last dose of study drug.
Time Frame: up to 152 days
Population: Safety Population: all participants who received at least 1 dose of study drug. Treatment groups for this population were determined according to the actual treatment the participant received on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 37 | 36 | 35 | 37
Participants | 20 | 20 | 25 | 28

5. Secondary Outcome: PC Period: Number of Participants With Any ≥Grade 3 TEAE
Description: A TEAE is any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug up to 30 days after the last dose of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events version 5.0 Grades 1 through 5. The investigator made an assessment of intensity for each AE and serious adverse event (SAE) reported during the study and assigned it to 1 of the following categories. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 152 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 37 | 36 | 35 | 37
Participants | 0 | 1 | 1 | 2

6. Secondary Outcome: Extension Period: Number of Participants With Any TEAE
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE is any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug up to 30 days after the last dose of study drug.
Time Frame: up to 215 days
Population: Extension Evaluable Population: all participants who received at least 1 dose of povorcitinib during the Extension Period
Measure: Count of Participants; unit: Participants
Groups:
- Placebo to Povorcitinib 45 mg: Participants who received placebo during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch Numerical Rating Scale (NRS) score and Investigator's Global Assessment-Treatment Success (IGA-TS) who did not receive rescue therapy during the placebo-controlled period.
- Povorcitinib 15 mg to 45 mg: Participants who received povorcitinib 15 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Povorcitinib 45 mg: Participants who received povorcitinib 45 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for an additional 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Povorcitinib 75 mg to 45 mg: Participants who received povorcitinib 75 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Placebo to Povorcitinib 75 mg: Participants who received placebo during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Povorcitinib 15 mg to 75 mg: Participants who received povorcitinib 15 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Povorcitinib 45 mg to 75 mg: Participants who received povorcitinib 45 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
- Povorcitinib 75 mg: Participants who received povorcitinib 75 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for an additional 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
Arm/Group | Placebo to Povorcitinib 45 mg | Povorcitinib 15 mg to 45 mg | Povorcitinib 45 mg | Povorcitinib 75 mg to 45 mg | Placebo to Povorcitinib 75 mg | Povorcitinib 15 mg to 75 mg | Povorcitinib 45 mg to 75 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 1 | 4 | 8 | 15 | 30 | 25 | 23 | 18
Participants | 0 | 3 | 5 | 7 | 20 | 19 | 16 | 13

7. Secondary Outcome: Extension Period: Number of Participants With Any ≥Grade 3 TEAE
Description: as for outcome 5
Time Frame: up to 215 days
Population: Extension Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to Povorcitinib 45 mg | Povorcitinib 15 mg to 45 mg | Povorcitinib 45 mg | Povorcitinib 75 mg to 45 mg | Placebo to Povorcitinib 75 mg | Povorcitinib 15 mg to 75 mg | Povorcitinib 45 mg to 75 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 1 | 4 | 8 | 15 | 30 | 25 | 23 | 18
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last dose of study drug (up to approximately 44 weeks)
Description: Adverse events have been reported for members of the Safety Population, comprised of all participants who received at least 1 dose of study drug.
Groups:
- Povorcitinib 45 mg to 45 mg: Participants who received povorcitinib 45 mg during the 16-week placebo-controlled period and were classified as responders at Week 16 received povorcitinib 45 mg QD for an additional 24 weeks in the extension period. Responders were defined as participants who had a ≥4-point decrease in Itch NRS score and IGA-TS who did not receive rescue therapy during the placebo-controlled period.
- Povorcitinib 75 mg to 75 mg: Participants who received povorcitinib 75 mg during the 16-week placebo-controlled period and were classified as non-responders at Week 16 received povorcitinib 75 mg QD for an additional 24 weeks in the extension period. Non-responders were defined as participants not meeting the definition of a responder.
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg | Placebo to Povorcitinib 45 mg | Povorcitinib 15 mg to 45 mg | Povorcitinib 45 mg to 45 mg | Povorcitinib 75 mg to 45 mg | Placebo to Povorcitinib 75 mg | Povorcitinib 15 mg to 75 mg | Povorcitinib 45 mg to 75 mg | Povorcitinib 75 mg to 75 mg
All-Cause Mortality (participants affected / at risk) | 0/37 | 1/36 | 0/35 | 0/37 | 0/1 | 0/4 | 0/8 | 0/15 | 0/30 | 0/25 | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/37 | 2/36 | 4/35 | 3/37 | 0/1 | 0/4 | 0/8 | 1/15 | 0/30 | 1/25 | 2/23 | 3/18
Other Adverse Events (participants affected / at risk) | 14/37 | 17/36 | 19/35 | 22/37 | 0/1 | 3/4 | 5/8 | 6/15 | 15/30 | 15/25 | 13/23 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | Povorcitinib 15 mg (N=36) | Povorcitinib 45 mg (N=35) | Povorcitinib 75 mg (N=37) | Placebo to Povorcitinib 45 mg (N=1) | Povorcitinib 15 mg to 45 mg (N=4) | Povorcitinib 45 mg to 45 mg (N=8) | Povorcitinib 75 mg to 45 mg (N=15) | Placebo to Povorcitinib 75 mg (N=30) | Povorcitinib 15 mg to 75 mg (N=25) | Povorcitinib 45 mg to 75 mg (N=23) | Povorcitinib 75 mg to 75 mg (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | Povorcitinib 15 mg (N=36) | Povorcitinib 45 mg (N=35) | Povorcitinib 75 mg (N=37) | Placebo to Povorcitinib 45 mg (N=1) | Povorcitinib 15 mg to 45 mg (N=4) | Povorcitinib 45 mg to 45 mg (N=8) | Povorcitinib 75 mg to 45 mg (N=15) | Placebo to Povorcitinib 75 mg (N=30) | Povorcitinib 15 mg to 75 mg (N=25) | Povorcitinib 45 mg to 75 mg (N=23) | Povorcitinib 75 mg to 75 mg (N=18)
Aspergillus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (7) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 6 (7) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint capsule rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen myxoedematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 2 (4) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT05061693/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT05061693/SAP_001.pdf